CLINICAL TRIAL: NCT00526409
Title: LAL-AR-N-2005: Study Treatment for Children High Risk Acute Lymphoblastic Leukemia
Brief Title: LAL-AR-N-2005:Study Treatment for Children High Risk Acute Lymphoblastic Leukemia
Acronym: LAL-AR-N-2005
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-AR-N-2005
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Prednisolone; Daunorubicin; Vincristine; Asparaginase; Cyclophosphamide; Methotrexate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Prednisolone — Induction: 60 mg/m2/day, oral or i.v x 21 days and 30 mg/m2/day oral or iv x 7 days Reinduction-Intensification Treatment: 60 mg/m2/d x 14 days and 30 mg/m2/day oral x 7 days
Drug: Daunorubicin — Induction: 30 mg/m2, i.v, days 1, 8, 15, 22 Consolidation (Bloc II)30 mg/m2, i.v, day 1
Drug: Vincristine — Induction: 1,5 mg/m2 iv, days 1, 8, 15, 22 Consolidation (Bloc I):1,5 mg/m2 iv, days 1, 8 Consolidation (Bloc II):1,5 mg/m2 iv, days 1, 8 Reinduction: 1,5 mg/m2 iv, days 1, 8 Maintenance:1,5 mg/m2 iv, day 22
Drug: L-Asparaginase — Induction: 10.000 U/m2 im or iv, days 9,11,13,16,18,20,23,25,27 Consolidation (Bloc II): 20.000 U/m2 im or iv, day 7 Maintenance: 20.000 U/m2 im or iv, day 22
Drug: Cyclophosphamide — Induction: 500 mg/m2 iv, days 1, 2, 29 Consolidation (Bloc I): 500 mg/m2 iv, day 8 Reinduction:500 mg/m2 iv, day 15
Drug: Methotrexate — Consolidation (Bloc I): 5 g/m2 24 hours infusion Consolidation (Bloc II): 5 g/m2 24 hours infusion Reinduction: 3 g/m2 24 hours infusion Maintenance: 20 mg/m2/d, IM/week x 3 (1, 7, 14)
Drug: Cytosine Arabinoside — Consolidation (Bloc I): 1 g/m2/12 h iv, days 5, 6 Consolidation (Bloc II): 1 g/m2/12 h iv, days 5, 6 Reinduction: 1 g/m2/12 h iv, days 43, 44

SUMMARY:
The study objective is to improve the global results obtained with LAL-AR-93 study, reaching an event free survival between 60-70%.

Identify patients with bad prognosis, with minimal residual disease,who can benefit of allogenic bone marrow transplantation

DETAILED DESCRIPTION:
INDUCTION TREATMENT

Systemic chemotherapy:

PREDNISOLONE 60 mg/m2 /day, oral or i.v. x 21 days (1 to 22) 30 mg/m2 /day, oral or i.v. x 7 days (23 to 29)

DAUNORUBICIN 30 mg/m2 , i.v. days 1,8,15 and 22

VINCRISTINE 1,5 mg/m2, i.v. days 1,8,15 and 22

L-ASPARAGINASE 10.000U/m2 i.m or i.v day 9,11,13,16,18,20,23,25 and 27

CYCLOPHOSPHAMIDE 500 mg/m2 i.v. days 1,2 and 29

Intrathecal chemotherapy:

Days 1 and 22 according age:

Age <1 years 1-3 years >3 years

Methotrexate (MTX), mg 5 8 12 Ara-C, mg 16 20 30 Hydrocortisone,mg 10 10 20

Patients with <10% blasts in M.O (day 14), and in complete response on week 5 or 6, and without MDR, start consolidation-intensification phase.

Patients with >10% blasts in MO day +14 or without CR after induction treatment, start consolidation-intensification phase and identifier a donor for a transplantation.

CONSOLIDATION/INTENSIFICATION (C.I.)

Two sequential cycles, alternating bloc I and bloc II

BLOC I

DEXAMETHASONE 10 mg/m2/d vo. days 1 to 5 and 5 mg/m2/d vo. days 6 and 7

VINCRISTINE 1.5 mg/m2/d, i.v. days 1 and 8

METHOTREXATE 5 g/m2 24 hours infusion + AF, day 1

ARA-C 1 g/m2/12 h, i.v., days 5 and 6

MERCAPTOPURINE 100 mg/m2/d, oral, days 1 to 5

CYCLOPHOSPHAMIDE 500 mg/m2 i.v. el day +8

INTRATHECAL CHEMOTHERAPY day 1.

BLOC II

DEXAMETHASONE 10 mg/m2/d, v o. days 1-5 and 5 mg/m2/d, v o. days 6 and 7

VINCRISTINE 1.5 mg/m2/d, days 1 and 8

METHOTREXATE 5 g/m2 24 h infusion + AF, day 1

ARA-C 1 g/m2 i.v/12 h, days 5 and 6

DAUNORUBICINE 30 mg/m2 i.v.day 1

L-ASPARAGINASE 20.000 u/m2/d, i.m. or i.v. day 7

INTRATHECAL CHEMOTHERAPY day 1

Patients with CR and MRD negative, follow chemotherapy. Patients with MDR >0.01% after second cycle or considered previously MRD are candidates to allogenic transplantation after second cycle.

REINDUCTION/INTENSIFICATION TREATMENT (R.I.)

PREDNISOLONE 60 mg/m2/d, oral x 14 days (1-14) 30 mg/m2/d, oral x 7 days (15-22)

VINCRISTINE 1.5 mg/m2, i.v. x 2 days 1 and 8

DAUNORUBICINE 30 mg/m2 i.v x 2 , days 1 and 8

CYCLOPHOSPHAMIDE 500 mg/m2 I.V. day 15

-----------------------------------------

METHOTREXATE 3 g/m2 /24 h infusion + AF day 29

MERCAPTOPURINE 50 mg/m2/d, oral, days 29-35 and 43-50

ARA-C 1 g/m2/12 h., i.v., days 43 and 44

INTRATHECAL CHEMOTHERAPY , days 1, 15, 29 and 43

MAINTENANACE TREATMENT (M1)

Six cycles of:

MERCAPTOPURINE 50 mg/m2/d, oral x 21 days (1-21)

METHOTREXATE 20 mg/m2/d, i.m. /week x 3 (1,7,14)

PREDNISOLONE 60 mg/m2/d, oral x 7 days (22-28)

VINCRISTINE 1.5 mg/m2 i.v.day 22

ASPARAGINASE 20.000 u/m2 i.m. day 22

INTRATHECAL CHEMOTHERAPY day 22

MAINTENANCE TREATMENT (M2)

Diary mercaptopurine and weekly methotrexate at previous doses, until complete 24 months.

ELIGIBILITY:
Inclusion Criteria:

* High risk children with acute lymphoblastic leukemia

Exclusion Criteria:

* Mature B-ALL (FABL3)
* Mixed forms of ALL
* Patients with coronary disorders, valvular or hypertensive cardiopathy
* Patients with chronic liver disorders
* Chronic pulmonary disorders
* Renal insufficiency
* Neurologic disfunctions
* ECOG 3 and 4

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2005-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To improve the global results obtained in PETHEMA LAL-AR-93 study in terms of events free time | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bastida Pilar, Dr, Study Chair — Hospital Universitari Materno-Infantil Vall d'Hebron; Ribera Josep Mª, Dr, Study Chair — Germans Trias i Pujol Hospital
Locations (4):
- Spain (4):
  - Hospital materno Infantil vall d'Hebrón, Barcelona
  - Hospital Niño Jesús, Madrid
  - Hospital Infantil Carlos Haya, Málaga
  - Hospital Virgen de la Arrixaca, Murcia

REFERENCES:
- See also: Spanish association of Haematology — http://www.aehh.org